CLINICAL TRIAL: NCT04795193
Title: A Partially Randomized Patient Preference Trial to Assess the Quality of Life and Patency Rate After Minimally Invasive Cardiac Surgery-Coronary Artery Bypass Grafting: the MICS-CABG PRPP Trial
Brief Title: MInithoraCotomy vs Sternotomy for Multivessel Coronary Artery Bypass Grafting: A Partially Randomized Patient Preference Trial Assessing Quality of Life and Patency Outcomes
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MICS-CABG PRPP Trial
Record Dates: First submitted 2021-03-03; First posted 2021-03-12 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-08

CONDITIONS: Coronary Artery Bypass, Off-Pump; Minimally Invasive Cardiac Surgery
Keywords: Coronary Artery Bypass, Off-Pump; Minimally Invasive Surgical Procedures; Coronary Artery Bypass

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MICS-CABG (minithoractomy CABG) (Experimental): Patients undergoing MICS-CABG(minithoractomy CABG)
  Interventions: Procedure: Minimal invasive coronary surgery
- CABG (sterotomy CABG) (Active Comparator): Patients undergoing CABG (sterotomy CABG)
  Interventions: Procedure: Off-pump coronary artery bypass surgery

INTERVENTIONS:
Procedure: Minimal invasive coronary surgery — Off-pump multi-vessel coronary artery bypass grafting via left thoracotomy under minimally invasive conditions.
  Arms: MICS-CABG (minithoractomy CABG)
Procedure: Off-pump coronary artery bypass surgery — Off-pump multi-vessel coronary artery bypass grafting with conventional thoracotomy.
  Arms: CABG (sterotomy CABG)

SUMMARY:
This trial will address essential questions of the efficacy and safety of MICS-CABG in addition to the quality of life and patency rate of the grafts. The study will also address the impact of patients' preferences on external validity and internal validity. In this study, patients with a preference will be allocated to treatment strategies accordingly, whereas only those patients without a distinct preference will be randomized. The randomized trial is a 248-patient controlled, randomized, investigator-blinded trial. It is designed to compare whether treatment with MICS-CABG is beneficial in comparison to CABG. This study is aimed to establish the superiority hypothesis for the physical component summary (PCS) accompanied by the noninferiority hypothesis for overall graft patency. Patients with no treatment preference will be randomized in a 1:1 fashion to one of the two treatment arms. The primary efficacy endpoints are the PCS score at 30 days (1 month) after surgery and the overall patency rate of the grafts within 14 days ( before discharge) after surgery. Secondary outcome measures include the PCS score and patency rate at different time points. Safety endpoints include major adverse cardiac and cerebrovascular events, complications, bleeding, wound infection, death, etc.

DETAILED DESCRIPTION:
Objective and Hypothesis: The aim of this study is to investigate and compare the mid-term safety and efficacy end-points (SF-36 PCS at 30 days after surgery, etc.) in patients with complex coronary artery lesions (an indication of OPCAGB) who received MICS-CABG and those who received thoracotomy OPCABG. The investigators hypothesize that patients in MICS-CABG group have superior 1-month PCS score assessed by SF-36 post-surgery and noninferior postprocedural angiographic graft patency rate prior to discharge.

Intervention Methods:

1. MICS-CABG (experimental group): Off-pump multi-vessel coronary artery bypass grafting via left thoracotomy under minimally invasive conditions.

   1. Surgery preparation:

      General anesthesia, double lumen tracheal intubation. In the supine position, tilt 15° to the right. An automatic defibrillation electrode is attached to the right front and left rear chest wall, and the external defibrillator is connected. A small incision of 8-10 cm into the left anterior lateral 5th intercostal space was performed into the chest.
   2. Internal mammary artery acquisition:

      After entering the chest, the internal mammary artery (IMA) is exposed through a new minimal invasive retraction system. Single or bilateral IMA is obtained as needed. Separate the IMA From the middle segment (non-fat muscle coverage area) applied with an electric scalpel (15J), and the free range was up to the first rib to the fifth or sixth intercostal (IMA bifurcation).
   3. Bypass strategy:

      All procedures were performed under a non-cardiopulmonary situation, and vascular anastomosis was performed with the aid of a laparoscopic cardiac stabilizer. The stabilizer is smaller and does not occupy the operating space. The head of stabilizer can be rotated 360 degrees and the target vessel can be fixed at any angle. Bilateral internal mammary artery, radial artery and saphenous vein can be used as graft vessels. The bypass strategy is not particularly different from conventional bypass surgery, including aorta (AO)-saphenous vein graft (SVG) or radial artery (RA)-X1-X2-...( sequential anastomosis), left internal mammary artery (LIMA)-right internal mammary artery (RIMA) -RA or SVG(Y)-X, RIMA-left anterior descending (LAD), LIMA-RA or RIMA or SVG(I)-X1-X2 and so on.
   4. Vascular anastomosis:

      The target vessel is exposed through the pericardial suture, the heart is locally fixed with the aid of a cardiac stabilizer, and the target vessel is inserted shunt to avoid hemodynamic disorder and arrhythmia. Vascular anastomosis is performed by 8-0 polypropylene suture.
   5. Aortic exposure and proximal anastomosis:

   Place gauze behind the aorta, expose the aorta with the right pericardial suspension suture, temporary block aortic anterior wall with a soft-chain sidewall clamp, Punch on the aortic anterior wall with 3.5 mm puncher, anastomose SVG or RA on AO with 6-0 polypropylene suture.
2. OPCABG (control group): Off-pump multi-vessel coronary artery bypass grafting with conventional thoracotomy.

Randomization Procedure:

Eligible patients will be randomized to MICS-CABG or OPCABG group with an allocation ratio of 1:1 after providing written informed consent. The randomization sequence will be generated by an independent statistician with block randomization method (block size=4 or 6). Each enrolled patient will be allocated to MICS-CABG or OPCABG group within 24-48 hours prior to surgery in the order of the assigned number in the allocation table uploaded in the electronic data capture (EDC) system. The allocation table will be concealed from researchers during research process.

Patient Selection:

Details are shown in the Eligibility Criteria part.

Measurements:

1. Baseline Measurements:

   1. General Information: sex, age, body mass index.
   2. Medical History and Comorbidity: smoking status, history of diabetes (oral hypoglycemic agents, insulin therapy, HbA1c greater than 7.0%, postprandial blood glucose greater than 11.1 mmol/L, fasting plasma glucose greater than 7.0 mmol/L), previous stroke, hyperlipidemia (under drug therapy, serum cholesterol greater than 5.72 mmol/L or triglyceride greater than 1.7 mmol/L at admission), hypertension (blood pressure greater than 140/90 mmHg without medication), renal insufficiency (dialysis or serum creatinine level greater than 140 mmol/L or creatinine clearance rate less than 30 mL/min), peripheral vascular disease [preoperative ultrasound or computed tomography (CT) confirmed peripheral vascular stenosis greater than 50%], previous history of cardiac surgery, previous percutaneous coronary intervention (PCI) history (balloon dilatation or stent implantation), previous myocardial infarction (MI) [pathological Q wave on ECG, definite evidence of elevation of creatine kinase (CK-MB) or troponin (cTnI) greater than 10 times of normal value with st-t segment elevation on cardiogram].
   3. Preoperative Status: SF-36, Seattle angina questionnaire (SAQ) score, classification of angina (stable angina pectoris, unstable angina pectoris, non st-t segment elevation myocardial infarction, st-t segment elevation myocardial infarction), New York Heart Association (NYHA) heart function classification, severe pulmonary insufficiency [post-bronchodilator forced expiratory volume in 1 s (FEV1)/forced vital capacity (FVC)<70% and FEV1%predicted<50% or partial pressure of oxygen (pO2)<60 mmHg or partial pressure of carbon dioxide (pCO2)>40 mmHg without oxygen therapy].
   4. Preoperative Examination: creatinine (Cr), N-terminal pro brain natriuretic peptide (NT-proBNP), preoperative cardiac function [ejection fraction (EF)%, left ventricular end-diastolic myocardial mass (LVEDm)], SYNTAX score (evaluated by two cardiologist).
   5. Preoperative Medication (within 1 week): aspirin, P2Y12 receptor antagonist (clopidogrel, ticagrelor), glycoprotein IIb/IIIa inhibitor (abciximab, eptifibatide, tirofiban, etc.).
2. Outcomes: Details are shown in the Outcome Measures part.

Follow-ups:

Patients will be followed at 7 days, 14 days, 30 days (1 month), 3 months, 6 months, and 12 months after surgery.

Sample Size:

1. Superiority Hypothesis:

   Objective: To establish the superiority hypothesis for PCS (Physical Component Score).

   Margin of Superiority: Set at 2, based on clinically and statistically significant differences, ethical considerations, cost, and feasibility.

   Assumptions:

   Difference between groups: 7. Estimated standard deviation: 10. Confidence interval: Two-sided 95%. Power: 90%. Calculated Sample Size: 172 patients (86 per group). Dropout Rate: Anticipated at 10%. Total Sample Size Required: 190 patients (95 per group).
2. Non-Inferiority Hypothesis:

   Objective: To establish the non-inferiority hypothesis for the overall patency rate of grafts.

   Margin of Non-Inferiority: Set at 6%.

   Assumptions:

   Expected overall patency rate: 96% in both MICS-CABG and sternotomy CABG. Power: 90%. Type 1 error: One-sided, 2.5%. Reduction in MICS-CABG: 0%. Calculated Sample Size: 496 grafts (248 per group). Dropout Rate: Allows for 10% loss to follow-up. Patients Required: Based on an average of at least 2 grafts per patient, a sample size of 248 patients (124 per group) is necessary.

   Total Sample Size Required: 248 patients with equal allocation to two arms.
3. Summary:

Totally, 248 patients ensure adequate power for both hypotheses.

Statistical Analysis:

The primary endpoint is SF-36 PCS at 30 days and graft patency after surgery. The analysis on the primary endpoint will be conducted according to the basic principle of ITT.

For baseline characteristics, mean and standard deviation will be described for continuous data with normal distribution, while median and interquartile range (IQR) will be used to depict continuous skewed data. Frequencies and percentages will be demonstrated for categorical variables. For group comparisons, t-test will be used for normal distributed variables, Mann-Whitney U test will be applied for skewed variables, while Pearson's chi-squared test or Fisher's exact test will be conducted for categorical variables.

For the primary endpoint: For the PCS score superiority test will be adopted, while for the patency rate of the graft, non-inferiority test will be used.

For secondary endpoints, t-test will be used for normal distributed variables, Mann-Whitney U test will be applied for skewed variables, while Pearson's chi-squared test or Fisher's exact test will be conducted for categorical variables. Survival analysis will be applied for time-to-event data [time to the first major adverse cardiovascular and cerebrovascular events (MACCE) within1, 3, 6, 12 ,36 and 60 months after surgery].

Statistical significance is defined as the two-sided p-value less than 0.05. All analyses were performed using Statistical Package for the Social Sciences (SPSS) version 26.0 or Statistical Analysis System (SAS) version 9.4 or later.

ELIGIBILITY:
Inclusion Criteria:(A patient will be included in the study when the following criteria and requirements are met)

① Patient age of ≥25 years but ≤85 years, and patients with CAD who require multivessel coronary bypass surgery. ② Angina that affects daily life and work and is uncontrollable with conservative treatment. ③ Significant stenosis in the left main (LM) coronary artery, left anterior descending (LAD) branch or left circumflex (LCX) branch >70%. ④ Severe stenosis (stenosis degree >70%) of three main branches of the coronary artery (anterior descending branch, circumflex branch, right coronary artery) with the need to undergo off-pump coronary artery bypass surgery.

Exclusion Criteria:

* Unstable preoperative hemodynamic status requiring emergency surgery
* Severe emphysema, hypoxemia [post-bronchodilator forced expiratory volume in 1 s (FEV1)/forced vital capacity (FVC)<70% and FEV1%predicted<50% or partial pressure of oxygen (pO2)<60 mmHg or partial pressure of carbon dioxide (pCO2)>40 mmHg without oxygen therapy]
* Old large area myocardial infarction, no viable myocardium based on isotope and echocardiography examination, significant cardiac enlargement, cardiothoracic ratio>0.75, EF<30%, left ventricular diastolic diameter (LVDd)>60 mm, left ventricular aneurysm or severe arrhythmia, prone to experience unstable preoperative hemodynamic status during surgery
* Severe pleural adhesion, chest deformity, or previous thoracic radiotherapy
* Previous open heart surgery
* Simultaneous valve or other cardiac surgery
* Planned cardiopulmonary bypass surgery
* Poor condition of myocardial infarction (MI), extensive lesion, distal or entire diffuse stenosis, or inability to match lumen due to small diameter (<1.0 mm) or severe calcification
* Others: Terminal cancer, uncontrolled infection, bleeding, progressive degenerative systemic disease, severe brain injury, multiple organ failure and other major organ dysfunction such as severe liver dysfunction, severe heart failure or cardiogenic shock, intolerance to surgery, and other contraindications of CABG

Ages: 25 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Estimated)
Dates: Start 2021-04-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
SF-36 PCS score (Physical component summary of medical outcomes study-short form 36-item scores) at 30 days (1month) after surgery | 30 days (1 month) after surgery
  The SF-36 is a concise health test that features Physical Functioning (PF), Roe-Physical (RP), Bodily Pain, General Health (GH), Vitality (VT), Social Functioning (SF), Roe-Emotional (Emotional) and Mental Health (MH) functioning and comprehensively summarizes the quality of life of the respondents across 8 aspects. The PCS and mental component summary (MCS) can be calculated from the eight abovementioned indicators with different weights. The PCS and the MCS each range from 0 to 50, with a lower score indicating worse quality of life (QoL) and a higher score indicating better QoL.
Overall patency rate of the grafts | within 14 days after surgery (before discharge)
  the patency rates of the LIMA, RIMA, saphenous vein graft (SVG) and radial artery (RA) will be evaluated by the Fitzgibbon A+B grade

SECONDARY OUTCOMES:
Perioperative transfusion volume | Intraoperative and 14 days after surgery
  Perioperative transfusion number (U) of red blood cell
Incidence of cardiopulmonary bypass conversion | 14 days after surgery
  Perioperative incidence of cardiopulmonary bypass conversion
Percentage of intra-aortic balloon pump (IABP) and extracorporeal membrane oxygenation (ECMO) usage | 14 days after surgery
  Perioperative percentage of IABP and ECMO usage
Incidence of secondary surgery | 14 days after surgery
  All cause secondary surgery event such as bleeding, hemodynamic instability, sternum fracture or wound infection, etc.
Incidence of adverse events of wound healing | 14 days, 1 month, 3 months, 6 months and 12 months after surgery
  Adverse events of wound healing include redness, exudation, cracking, delayed healing that need surgical suture
Incidence of perioperative major adverse cardiovascular and cerebrovascular event (MACCE) | 30 days after surgery
  Major adverse cardiovascular and cerebrovascular event which is a composite endpoint of myocardial infarction, stroke and death
Incidence of atrial fibrillation | 30 days after surgery
  Perioperative incidence of atrial fibrillation
Incidence of renal failure | 30 days after surgery
  Perioperative incidence of renal failure
Incidence of re-intubation | 14 days after surgery
  Perioperative incidence of re-intubation
Length of stay after surgery (days) | 14 days after surgery
  Perioperative number of days staying in hospitals after surgery
Intensive care unit (ICU) duration after surgery (hours) | 14 days after surgery
  Perioperative duration of ICU stay after surgery
Duration of mechanical ventilation application (hours) | 14 days after surgery
  Perioperative duration of mechanical ventilation application
Physical limitation score of Seattle angina questionnaire (SAQ) | 1 month, 3 months, 6 months and 12 months after surgery
  The SAQ quantifies 5 domains measuring the impact of angina on patients' health status: physical limitation (9 items), angina stability (1 item), angina frequency (2 items), treatment satisfaction (4 items), and disease perception (3 items). Each scale is transformed to a score of 0 to 100, where higher scores indicate better function.
Angina stability score of Seattle angina questionnaire (SAQ) | 1 month, 3 months, 6 months and 12 months after surgery
  The SAQ quantifies 5 domains measuring the impact of angina on patients' health status: physical limitation (9 items), angina stability (1 item), angina frequency (2 items), treatment satisfaction (4 items), and disease perception (3 items). Each scale is transformed to a score of 0 to 100, where higher scores indicate better function.
Angina frequency score of Seattle angina questionnaire (SAQ) | 1 month, 3 months, 6 months and 12 months after surgery
  The SAQ quantifies 5 domains measuring the impact of angina on patients' health status: physical limitation (9 items), angina stability (1 item), angina frequency (2 items), treatment satisfaction (4 items), and disease perception (3 items). Each scale is transformed to a score of 0 to 100, where higher scores indicate better function.
Treatment satisfaction score of Seattle angina questionnaire (SAQ) | 1 month, 3 months, 6 months and 12 months after surgery
  The SAQ quantifies 5 domains measuring the impact of angina on patients' health status: physical limitation (9 items), angina stability (1 item), angina frequency (2 items), treatment satisfaction (4 items), and disease perception (3 items). Each scale is transformed to a score of 0 to 100, where higher scores indicate better function.
Disease perception score of Seattle angina questionnaire (SAQ) | 1 month, 3 months, 6 months and 12 months after surgery
  The SAQ quantifies 5 domains measuring the impact of angina on patients' health status: physical limitation (9 items), angina stability (1 item), angina frequency (2 items), treatment satisfaction (4 items), and disease perception (3 items). Each scale is transformed to a score of 0 to 100, where higher scores indicate better function.
Time to the first major adverse cardiovascular and cerebrovascular event (MACCE) after surgery | 1 month, 3 months, 6 months, 12 months, 36months and 60 months after surgery
  Major adverse cardiovascular and cerebrovascular event which is a composite endpoint of myocardial infarction, stroke and death
Incidence of readmission due to myocardial infarction (MI) | 1 month, 3 months, 6 months and 12 months after surgery
  Incidence of readmission due to MI during follow-ups
Incidence of readmission due to heart failure | 1 month, 3 months, 6 months and 12 months after surgery
  Incidence of readmission due to heart failure during follow-ups
Percentage of mid-term graft patency (evaluated by CT or angiography) | 12 months after surgery
  Percentage of mid-term graft patency evaluate by angiography or CT angiography
SF-36 PCS scores | 7-14 days (0.5 month) , 3 months, 6 months and 1 year after surgery
SF-36 MCS scores | 7-14 days, 1month, 3 months, 6 months and 1 year after surgery
Patency rate of the different material grafts | 14 days (before discharge) and 1 year after surgery
  the patency rates of the LIMA, RIMA, saphenous vein graft (SVG) and radial artery (RA) will be evaluated by the Fitzgibbon A+B grade
Bypass surgical variation index | within 7 days after surgery
  The actual graft number is compared with the preoperative strategy. If the actual number of grafts is less than that in the preoperative plan, the results will be recorded.
Intrahospital RBC transfusion volume | before discharge
  the amount of red blood cells (U) to be transfused during hospitalization.
Number of Participants with re-exploration for bleeding or other causes (not including wound-related causes) | within 1 year after surgery
  the requirement to return to the operating room for reopening of sternotomy or MICS CABG incision for any reason, such as bleeding, postoperative acute myocardial ischemia and unexplained circulatory instability. Debridement for DSWI or infection of anterior-lateral wounds will be excluded.
Wound infection rate | within 3 months after surgery
  wound dehiscence, effusion and secondary debridement and suture

CONTACTS AND LOCATIONS:
Overall Officials: Yunpeng Ling, Doctor, Study Chair — Peking University Third Hospital; Yichen Gong, Doctor, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data that underlie the results (text, tables, figures, and appendices) reported in the publication of summary data, study protocol, statistical analysis plan (SAP), analytic code will be shared from 6 months to 3 years following article publication. All above could be shared with researches who provide a methodologically sound and feasible proposal approved by principal investigator (email address: yunpengling@163.com) and a signed data access agreement.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: From 6 months to 3 years following the article publication of summary data.
Access Criteria: Researches should send a proposal to yunpengling@163.com or 18611693463@126.com. If the proposal is methodologically sound, feasible and approved by the principal investigator, data requestor could gain access after signing a data access agreement.